CLINICAL TRIAL: NCT00762853
Title: Development of Clinical Method to Triclosan Retention in Plaque Following Brushing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2008-PLA-16-RR
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2010-08

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): fluoride toothpaste from Thailand
  Interventions: Drug: Fluoride
- B (Active Comparator): fluoride/triclosan/copolymer toothpaste
  Interventions: Drug: Fluoride and triclosan

INTERVENTIONS:
Drug: Fluoride — Brush half mouth once with assigned study treatment
  Arms: A
Drug: Fluoride and triclosan — Brush half mouth once with assigned study treatment
  Other Names: Colgate Total toothpaste
  Arms: B

SUMMARY:
The objective is to develop a method to determine active ingredient uptake in oral care products.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteer 18 - 65 years of age (inclusive).
* Good general health with a minimum of twenty (20) natural, uncrowned teeth (excluding third molars)
* Able and willing to sign the informed consent form.
* Plaque score of at least 1.5 on the modified Quigley-Hein plaque index.
* No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental procedures/visits
* Medical condition which precludes not eating/drinking for 2 hours
* Advanced periodontal disease (gum disease)
* 5 or more decayed, untreated dental sites (cavities)
* Diseases of the soft or hard oral tissues
* Orthodontic appliances
* Abnormal salivary function
* Use of drugs that can affect salivary flow
* Use of antibiotics one (1) month prior to or during this study
* Use of any over the counter medications other than analgesics (i.e. aspirin, ibuprofen, acetaminophen, naproxyn, etc)
* Pregnant or breastfeeding.
* Participation in another clinical study in the month preceding this study
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triantana, DDS, Principal Investigator
Locations (1):
- Mahidol University, Bangkok, Bangkok 10110, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: Subjects were screened for medical and oral health criteria and then began a 1 week washout period with fluoride toothpaste.
Groups:
- Placebo First, Active Second: subjects brushed their teeth with Fluoride toothpaste (Placebo) during the first intervention, then brushed with the fluoride/triclosan (Active) toothpaste during the second intervention.
- Active Toothpaste First, Then Placebo: Subjects brushed their teeth with the fluoride/triclosan(Active) toothpaste during the first intervention, then brushed with the fluoride alone toothpaste(placebo) during the second intervention.
Period: First Treatment Period
Arm/Group | Placebo First, Active Second | Active Toothpaste First, Then Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: 1 Week Washout After Treatment 1
Arm/Group | Placebo First, Active Second | Active Toothpaste First, Then Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | Placebo First, Active Second | Active Toothpaste First, Then Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Active Second | Active Toothpaste First, Then Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.9) | 35.6 (9.9) | 35.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Thailand | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Triclosan Concentration in Dental Plaque
Description: Triclosan is analyzed by gas chromatography (GC) with Atomic Emission Detection (480 nm) and quantitated by determining the ration of the peak height of triclosan to the peak height of an internal standard and relating the result to corresponding ratios of calibration standards.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ppm levels of triclosan
Groups:
- Fluoride Toothpaste (Placebo): fluoride only toothpaste
- Active Toothpaste: fluoride/triclosan/copolymer(Active) toothpaste
Arm/Group | Fluoride Toothpaste (Placebo) | Active Toothpaste
Number analyzed (Participants) | 20 | 20
ppm levels of triclosan | 0 (0) | 1.8 (1.2)
Statistical Analysis 1: Comparison: Fluoride Toothpaste (Placebo) vs Active Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 16 days
Arm/Group | Placebo First, Active Second | Active Toothpaste First, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less